CLINICAL TRIAL: NCT00450840
Title: Simvastatin in Patients With Septic Shock
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3732006
Record Dates: First submitted 2007-03-21; First posted 2007-03-22 (Estimated); Last update posted 2007-09-17 (Estimated); Status verified 2007-09

CONDITIONS: Septic Shock
Keywords: septic shock; simvastatin
MeSH Terms: conditions — Shock, Septic | interventions — Simvastatin

INTERVENTIONS:
Drug: Simvastatin

SUMMARY:
The beneficial effect of statins to prevent cardiovascular events in patients at risk is well established. Recent trials demonstrated that statins can exert a number of vascular actions independent of lipid lowering. Short-term simvastatin therapy recently has been reported to reduce mortality in 2 different animal models of sepsis. Pleiner and coworkers could demonstrate potent vasoprotective properties of simvastatin during Escherichia coli endotoxin induced endotoxemia in healthy volunteers. In a population-based cohort analysis it was demonstrated that administration of statins was associated with a reduced risk of subsequent sepsis. Thus, simvastatin treatment may offer a new therapeutic strategy for clinical conditions associated with inflammation like severe sepsis and septic shock. The aim of the present study is to test the hypothesis that short term treatment with simvastatin may mitigate the detrimental vascular effects of acute inflammation in patients admitted to the intensive care unit requiring treatment for septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Septic Shock for less than 48 hours

Exclusion Criteria:

* Pregnancy
* Unable to receive enteral medications
* Expected survival of less than 72 hours
* Treatment in the previous 3 weeks with simvastatin or other HMG-CoA reductase inhibitors
* History of hypersensitivity to the trial drug or to drugs with a similar chemical structure
* History of known or suspected porphyria
* High risk of rhabdomyolysis (multiple trauma, crush injuries, extensive burns, baseline creatinine kinase (CK) ≥ten-times upper limit of normal
* Hemorrhagic shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Time to shock reversal as defined by cessation of vasopressor support > 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schenk, MD, Principal Investigator — Medical University of Vienna, Intensive Care Unit
Locations (1):
- Medical University of Vienna, Dep. of Internal Medicine III, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Dobesh PP, Olsen KM. Statins role in the prevention and treatment of sepsis. Pharmacol Res. 2014 Oct;88:31-40. doi: 10.1016/j.phrs.2014.04.010. Epub 2014 May 2. PMID 24794878